CLINICAL TRIAL: NCT06013293
Title: Evalution of Postoperative Pain With Resin Based Sealer vs Zinc Oxide Eugenol Sealer After Single Visit Endodontic
Brief Title: Evaluation of Postoperative Pain With Resin Based Sealer vs Zinc Oxide Eugenol Based Sealer After Single Visit Endodontic
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Pakistan Institute of Medical Sciences (Other Government)
Responsible Party: Principal Investigator, Ahsen amin, Principal investigator, Pakistan Institute of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SOD/ERB/2023/19
Record Dates: First submitted 2023-08-22; First posted 2023-08-28 (Actual); Last update posted 2023-08-28 (Actual); Status verified 2023-08

CONDITIONS: Post Operative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — epoxy resin-based root canal sealer

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Zinc oxide eugenol based sealer (Experimental): Root canal treatment will be performed in posterior teeth.In this group the root canal will be dried with paper points and obturated with using gutta-percha cones and zinc oxide eugenol sealer. Coronal access cavities will be restored with direct composite restorations using dentinal adhesives and universal composite resin . Postoperative VAS scores will be recorded after 24 h and 48 h to determine their post-operative pain.
  Interventions: Procedure: Zinc oxide eugeonal based sealer
- Resin based sealer (Active Comparator): Root canal treatment will be performed in posterior teeth.In this group the root canal will be dried with paper points and obturated with using gutta-percha cones and resin based sealer. Coronal access cavities will be restored with direct composite restorations using dentinal adhesives and universal composite resin . Postoperative VAS scores will be recorded after 24 h and 48 h to determine their post-operative pain.
  Interventions: Procedure: Resin Based Sealer

INTERVENTIONS:
Procedure: Zinc oxide eugeonal based sealer — Zinc oxide-eugenol (ZOE)- based preparations, which have been used in root canal obturation (RCO) for over a hundered years and are known for their antimicrobial activities.slight microleakage and zinc oxide-eugenol's superior antibacterial property,slight microleakage and concerning the lower cytotoxicity, the zinc oxide-eugenol (ZOE) sealer can be used for root canal obturation as an endodontic sealer.After root canal prepartion , the root canal will be dried with paper points and obturated using gutta-percha cones and zinc oxide eugenol sealer.
  Arms: Zinc oxide eugenol based sealer
Procedure: Resin Based Sealer — resin-based sealer used frequently as a gold standard for endodontic sealers, due to its good physicochemical properties and provide satisfactory adhesion interface with dentin radicular surface.After root canal preparation, the root canal will be dried with paper points and obturated using gutta-percha cones and Resin based sealer
  Arms: Resin based sealer

SUMMARY:
The goal of root canal therapy is thorough disinfection and obturation of the root canal system in all its dimensions and promote periradicular tissue repair.This study was done to compare the postopertaive pain after single visit endodontics using resin based sealer and zinc oxide eugeonal sealer

DETAILED DESCRIPTION:
A total of 100 patients requiring endodontic treatment for permanent molar in accordance with the inclusion and exclusion criteria will be selected for the study. The treatment and study design will be explained to the patients in their own comprehendible language and a written informed consent will be obtained from the voluntary patients who participated in the study. A cold test and electric pulp-test was used to assess pulp vitality. Based on clinical and radiographic findings, the patients diagnosis of irreversible pulpitis. Patients will be randomly divided into two groups Group A = resin based sealer and Group B = Zinc oxide eugenol sealer. Prior to treatment the patients will be instructed how to complete a visual analog scale (VAS) to determine their pain score. The VAS included a 10 cm straight horizontal line numbered at each centimeter with the following criteria.Local anesthetic with 2% lignocaine containi Local anesthetic with 2% lignocaine containing 1:80000 epinephrine will be administered to each patient after recording preoperative pain levels . A rubber dam will be applied. The endodontic access cavities will be prepared with endo access burs .Working length will be established with #10 K file and the root canal will be instrumented with one shape rotary system up to #25.6% under copious irrigation with 3% sodium hypochlorite and normal saline. Before obturation root canals will be final rinse with 5 ml of 17% EDTA solution. In both groups, the root canal will be dried with paper points and obturated using gutta-percha cones and Resin based sealer/zinc oxide eugenol sealer. Coronal access cavities will be restored with direct composite restorations using dentinal adhesives and universal composite resin . Postoperative VAS scores will be recorded after 24 h and 48 h to determine their post-operative pain.

ELIGIBILITY:
Inclusion Criteria:

1. Patient who agree to participate in study
2. ASA CLASSIFICATION 1or 2
3. Minimum age of 18years old and maximum age of 65 years old
4. Maxillary and Mandibular single rooted teeth included in the study
5. Patient with symptomatic irreversible pulpitis with either normal apical tissue or symptomatic apical periodontitis.

Exclusion Criteria:

- 1. ASA Classification 3 to 5 2. Patient with immature apices and root resorption will be excluded from the study.

3. Severe periodontal problem. 4. Vertical or horizontal root fractures will be excluded from the study 5. Patients who will be already on analgesia within 24 hours excluded from study 6. Those requiring root canal treatment of two or more teeth ipsilaterally (since the pain caused by any of these teeth can result in false positive reading) will be excluded

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-08-30 (Estimated); Study Completion 2023-09-01 (Estimated)

PRIMARY OUTCOMES:
Post operative pain | immediately after the procedure
  . Postoperative Visual analogue pain scores will be recorded

CONTACTS AND LOCATIONS:
Locations (1):
- School of Dentistry, Islamabad, Pakistan